CLINICAL TRIAL: NCT04124198
Title: Quality of Life After Primary Transoral Robotic Surgery vs Intensity-modulated Radiotherapy for Patients With Early-stage Oropharyngeal Squamous Cell Carcinoma: A Randomized National Trial
Brief Title: Quality of Life After Primary TORS vs IMRT for Patients With Early-stage Oropharyngeal Squamous Cell Carcinoma
Acronym: QoLATI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian von Buchwald (Other)
Collaborators: Naestved Hospital (Other); Herlev Hospital (Other); Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Christian von Buchwald, Clinical Professor and Study Chair, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The QoLATI Study; DAHANCA 34 (Other: The Danish Head and Neck Cancer Group)
Record Dates: First submitted 2019-10-06; First posted 2019-10-11 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Oropharynx Cancer; Oropharynx Squamous Cell Carcinoma; Carcinoma, Squamous Cell; Carcinoma; Oropharyngeal Neoplasms; Neoplasms, Squamous Cell; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Pharyngeal Neoplasms Malignant and Unspecified; Otorhinolaryngologic Neoplasms; Head and Neck Neoplasms; Neoplasms by Site; Otorhinolaryngologic Diseases; Pharyngeal Diseases; Papillomavirus Infections; Virus Diseases; DNA Virus Infections; Tumor Virus Infections; Quality of Life
Keywords: Oropharyngeal squamous cell carcinoma T1-T2, N0-1; Transoral robotic surgery; Intensity Modulated Radiation Therapy
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Carcinoma; Neoplasms, Squamous Cell; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Otorhinolaryngologic Neoplasms; Head and Neck Neoplasms; Neoplasms by Site; Otorhinolaryngologic Diseases; Pharyngeal Diseases; Papillomavirus Infections; Virus Diseases; DNA Virus Infections; Tumor Virus Infections | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; Nimorazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transoral robotic surgery (TORS) (Experimental)
  Interventions: Procedure: Transoral Robotic Surgery (TORS) with neck dissection
- Intensity-Modulated Radiation Therapy (IMRT) (Active Comparator): Patients with clinical T1N0 stage are offered accelerated radiotherapy to 66 Gy/33fractions with concurrent nimorazole.
  Patients with clinical T2N0 stage are offered either accelerated radiotherapy to 66 Gy/33fractions with the option of weekly cisplatin to fit patients or hyper-fractionated accelerated radiotherapy to 76 Gy/56fractions both with concurrent nimorazole.
  Patients with clinical T1-T2, N1 stage are offered accelerated radiotherapy to 66 Gy/33 fractions and nimorazole with the addition of concurrent weekly cisplatin 40 mg/sqm to fit patients.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy (IMRT); Drug: Cisplatin; Drug: Nimorazole.

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy (IMRT) — Accelerated or hyper-fractionated radiotherapy
  Arms: Intensity-Modulated Radiation Therapy (IMRT)
Drug: Cisplatin — Concurrent weekly cisplatin 40 mg/sqm to fit patients
  Arms: Intensity-Modulated Radiation Therapy (IMRT)
Drug: Nimorazole. — Concurrent nimorazole
  Arms: Intensity-Modulated Radiation Therapy (IMRT)
Procedure: Transoral Robotic Surgery (TORS) with neck dissection — Robotic-assisted resection of the primary oropharyngeal tumour and ipsilateral selected neck dissection of lymph node levels II-IV. Patients with a primary base of tongue cancer or with significant involvement of tongue base or the soft palate defined as above 1 cm, will be offered a bilateral neck dissection of levels II-IV.
  Arms: Transoral robotic surgery (TORS)

SUMMARY:
Oropharyngeal squamous cell carcinoma (OPSCC) is now the most frequently diagnosed head and neck cancer in Denmark which is mainly due to the increase of Human Papillomavirus (HPV). Patients with HPV-positive OPSCC have a significantly higher survival rate compared to HPV-negative OPSCC. The traditional primary treatment modality in Denmark is Intensity Modulated Radiation Therapy (IMRT), and in advanced stages in combination with chemotherapy. Since 2009, Transoral Robotic Surgery (TORS) has enabled surgeons to perform minimally invasive surgery as an alternative to standard radiotherapy treatment which is considered the primary treatment for OPSCC in many countries. There is a lack of randomised trials comparing long-term functional outcomes after TORS or IMRT. Current data are mostly derived from retrospective studies with selection bias. However, several small retrospective studies have shown promising results when comparing the two treatment modalities in favour of TORS with regards to treatment related swallowing function and quality of life (QoL) without compromising survival outcomes.

This study aims to evaluate the early and long-term functional outcomes following two treatment arms 1) TORS combined with neck dissection and 2) IMRT±concurrent chemotherapy with a special focus on swallowing-related QoL.

DETAILED DESCRIPTION:
The current study is performed as a nationwide randomized phase III study that aims to investigate the long-term functional outcomes after primary TORS and neck dissection vs. IMRT±concurrent chemotherapy for early-stage oropharyngeal squamous cell carcinoma.

The study is a registered Danish Head and Neck Cancer Group (DAHANCA) 34 protocol.

The investigators hypothesise that primary TORS±adjuvant therapy will significantly improve the QoL at 12 months follow-up compared to IMRT±concurrent chemotherapy.

Primary endpoint: QoL measured by a composite MD Anderson Dysphagia Inventory (MDADI) score evaluated at 12 months follow-up after treatment (10-point difference)

Study design:

Patients who meet the inclusion criteria will be recruited from three Danish head and neck cancer centers: Copenhagen University Hospital Rigshospitalet, Aarhus University Hospital and Odense University Hospital.

Prior to treatment, all patients will be reviewed and examined at a multidisciplinary team conference.

Included patients will be randomized in 2:1 ratio:

Arm 1 (experimental), n=92 patients: TORS+neck dissection. Arm 2 (control), n=46 patients: IMRT±concurrent chemotherapy

DAHANCA Secretariat is responsible for the randomization key to either experimental or control arm. The investigators will stratify for p16, sex, tumour location and clinical tumor- and nodal-stage (T- and N-stage) classification at time of inclusion to avoid an uneven distribution in the experimental arm compared to the control arm.

Specifics for the experimental arm:

Patients with clinically positive neck (cN+) will be offered a staging neck within 8 days prior to the planned TORS. Based on final pathology of the neck specimen, patients will either be referred for definitive IMRT± concurrent chemotherapy (extracapsular extension (ECE), or more than two lymph node metastases) or they will undergo TORS (no extracapsular exension and maximally two lymph node metastases).

For patients with clinically no evidence of lymph node metastasis (cN0), neck dissection can be performed either before (within 8 days) or concurrently (same day procedure) with TORS.

Indications for adjuvant radiotherapy:

Nodal site:

* More than two lymph node metastases
* Two lymph node metastases and both above 1 cm in diameter.
* Any pathological positive lymph nodes (pN+) with extracapsular extension (ECE)
* A neck dissection nodal yield of less than 10 lymph nodes per side (after total embedding of the remaining fat tissue)

Tumour site:

* Involved or close resection margins of < 2 mm if free margins was not obtained after supplementary resections per-operatively or after re-resection in a secondary procedure.
* In case of stage migration to tumour stages T3 or T4, in an otherwise radical operation (R0), adjuvant therapy will be offered based on a postoperative consultation between the patient, the surgeon and an oncologist.

Indications for adjuvant chemotherapy:

• Insufficient resection margin (<2mm) or ECE

Specifics for the control arm:

Radiotherapy Quality Assurance Reviews are aimed to be performed before the third treatment fraction by a team from another head-neck oncology center consisting of one physicist and one oncologist. The patient specific review will address the following points according to the DAHANCA guideline: Clinical Target Volume (CTV) and Organs-at-Risk (OAR) delineation, target dose coverage, OAR dose sparing and treatment length.

Funding: The study protocol was initiated by the Department of Otorhinolaryngology, Head & Neck surgery at Copenhagen University Hospital Rigshospitalet. Funding grants have been received by the Danish Health Authority ("Midler til eksperimentel kræftkirurgi"), by the Copenhagen University Hospital Rigshospitalet ("Rammebevilling") and Odense University Hospital ("Forskningspulje mellem OUH og RH").

Data management and ethical considerations: Data is stored and handled in accordance with the Danish Data Agency regulations, The General Data Protection Regulation (GDPR) 2016/679 in European Union (EU) law on data protection and privacy for all individual citizens of the EU and the European Economic Area (EEA), and in compliance with the national data agreement between the study locations in compliance with the Danish Data Protection Agency approval (ID: RH-2017-362).

During the trial, the Good Clinical Practice (GCP) unit in Aarhus will monitor the study trial according to the given protocol and the current legislation. The monitoring period will consist of the first 12 months of inclusion until the primary endpoint.

This study has been approved by the Regional Committee on Health Research Ethics (ID: H-17031827)

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Able to provide informed consent
3. The Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status 0-2
4. Histologically confirmed oropharyngeal squamous cell carcinoma (exclusively palatine tonsils and base of tongue tumours) with known p16 status
5. Clinical tumour stage cT1-2 according to The Union for International Cancer Control (UICC), tumor (T), nodes (N), and metastases (M), (TNM) classification, 8th edition.
6. Clinical nodal stage cN0-1 according to UICC, TNM classification, 8th edition, however in p16 positive patients with unilateral metastasis, only a nodal metastasis up to a maximum of 4 cm in greatest diameter according to pre-operative imaging will be included.
7. Diagnostic imaging including computed tomography/magnetic resonance imaging (CT/MRI) performed within 14 days at time of randomization.
8. A tumour that is considered resectable according to MRI, clinical examination and/or ultrasound

Exclusion Criteria:

1. Serious medical comorbidities or ECOG/WHO performance status >2. Other contraindications to radiotherapy, chemotherapy or surgery
2. Inability to attend full course of radiotherapy or follow-up visits in the outpatient clinic
3. Distant metastasis
4. Clinically and radiologic signs of nodal extracapsular extension
5. Previous radiotherapy of the head and neck
6. Previous head and neck cancer
7. Significant trismus (maximum inter-incisal opening ≤ 35mm) [46]
8. Unable or unwilling to complete quality of life questionnaires
9. Posterior pharyngeal wall involvement
10. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Swallowing related quality of life by MDADI | evaluated at baseline, 3 and 12 months after treatment
  Difference in swallowing related quality of life measured by a composite MD Anderson Dysphagia Inventory (MDADI) score. The MDADI is a 20-item self-administered questionnaire that quantifies swallowing-related quality of life. Each item is scored on a 5 point Likert scale (strongly disagree, disagree, no opinion, agree, strongly agree). The composite MDADI score summarizes overall performance on remaining 19-items of the MDADI, as a weighted average of the physical, emotional, and functional subscale questions. Summary and subscale MDADI scores are normalized to range from 20 (extremely low functioning) to 100 (high functioning).

SECONDARY OUTCOMES:
Nasogastric or percutaneus tube dependency | evaluated at baseline, 3 and 12 months after treatment
  Tube dependency defined as number of days/weeks/months with tube inserted
Swallowing function by fiberendoscopic evaluation | evaluated at baseline, 3 and 12 months after treatment
  Fiberendoscopic Evaluation of Swallowing (FEES) is rated by following scales: a 8-point Penetration-Aspiration Scale (PAS) where a score of 1 reflects no entry of material into the airway, scores of 2-5 reflect penetration of material past the laryngeal additus into the supraglottic space and traveling as far as the true vocal folds, while scores of 6-8 reflect tracheal aspiration of material below the true vocal folds; Yale Pharyngeal Residue Severity Rating Scale: image-based assessment of post-swallow pharyngeal residue severity as observed during swallowing. Five-point ordinal rating scale based on residue location (vallecula and pyriform sinus) and amount (none, trace, mild, moderate, and severe); the summary DIGEST grading: grade 1= mild, grade 2= moderate, grade 3= severe, and grade 4= life threatening pharyngeal dysphagia.
Swallowing function by modified barium swallowing | evaluated at baseline, 3 and 12 months after treatment
  Modified Barium Swallowing (MBS) is a fluoroscopic procedure designed to determine whether food or liquid is aspirated. Following scales are used to assess MBS: a 8-point Penetration-Aspiration Scale (PAS): a score of 1 reflects no entry of material into the airway, scores of 2-5 reflect penetration of material past the laryngeal additus into the supraglottic space and traveling as far as the true vocal folds, while scores of 6-8 reflect tracheal aspiration of material below the true vocal folds; the summary DIGEST grading: grade 1= mild, grade 2= moderate, grade 3= severe, and grade 4= life threatening pharyngeal dysphagia.
Patient reported quality of life by EORTC-QLQ-H&N35 | evaluated at baseline, 3 and 12 months after treatment
  Measured by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaires EORTC-QLQ-H&N35. The head and neck-specific module EORTC QLQ-H&N35 contains 35 items, which can be condensed into 7 multi-item and 11 single-item scales. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Patient reported quality of life by EORTC QLQ-C30 | evaluated at baseline, 3 and 12 months after treatment
  Measured by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire EORTC QLQ-C30. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Treatment-related pain | evaluated at baseline up to 12 months after treatment
  Daily (experimental arm) or weekly (control arm) self-reported visual analogue scale (VAS) score from 0-10 points in which a higher score indicates greater pain intensity. Measured until no treatment-related pain is recorded by the patient and with no need of treatment-related pain medication
Weight | evaluated at baseline, 3 and 12 months after treatment
Patients returning to work after treatment | evaluated at baseline, 3 and 12 months after treatment
  Defined as the time (number of days) before returning to work or failure to do so after treatment.
Morbidity after staging neck after staging neck dissection | evaluated from time of neck dissection up to 14 days after treatment
  Monitoring of events of bleeding, lymphedema or impaired nerve function after staging neck dissection
Nerve function | evaluated at baseline and up to 12 months after treatment
  Evaluation of nerve function at risk during surgery (spinal accessory, hypoglossal, marginal mandibular branch of the facial nerve, lingual and vagal nerve) will be assessed by a clinical examination based on the innervation and function of each nerve during follow-up after surgery. Nerve function is determined as dichotomous variable: functioning/not-functioning.
Late toxicity | evaluated at 3, 6, 12, 24, 36, 48 and 60 months after treatment
  Using The Radiation Therapy Oncology Group/The European Organization for Research and Treatment of Cancer (RTOG/EORTC) Late Radiation Morbidity Score. Uses a grading system from 0-5 for different tissue organs: 0 - no symptoms, 5 - death directly related to radiation effects
Overall survival | evaluated from time of randomization up to 5 years
  Time from randomization to death from any cause.
Disease-free survival | evaluated from time of randomization up to 5 years
  Time from randomization to sign of cancer is found.
Disease-specific survival | evaluated from time of randomization up to 5 years
  Time from randomization to death from the disease (oropharyngeal cancer).
Distant recurrence | evaluated from time of randomization up to 5 years
  Time from randomization to distant recurrence
Loco-regional recurrence | evaluated from time of randomization up to 5 years
  Time from randomization to recurrence in same T-site or N-site as initial cancer localization

CONTACTS AND LOCATIONS:
Overall Officials: Christian von Buchwald, MD, DMSc., Study Chair — Department of Otorhinolaryngology, Head and Neck Surgery, Copenhagen University Hospital Rigshospitalet; Niclas Rubek, MD, Principal Investigator — Department of Otorhinolaryngology, Head and Neck Surgery, Copenhagen University Hospital Rigshospitalet
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-12-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT04124198/SAP_000.pdf